CLINICAL TRIAL: NCT04585100
Title: Phase 1/2a, Randomized, Double-Masked, Placebo-Controlled, Multi-center Study Assessing the Safety, Tolerability, And Efficacy Of FM101 In Patients With Ocular Hypertension, And To Assess The Relative Bioavailability Of The FM101 Oral Tablet Formulation In Healthy Participants
Brief Title: FM101 Safety, Tolerability, Efficacy Study in the Patients With Ocular Hypertension
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Future Medicine (Industry)
Collaborators: Futuremedicine Australia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: FM101-CTP2-002
Record Dates: First submitted 2020-09-07; First posted 2020-10-14 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-12

CONDITIONS: Ocular Hypertension
Keywords: Ocular Hypertension; OHT; FM101
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioequivalent test of FM101 oral solution and FM101 tablet (Experimental)
  Interventions: Drug: FM101 tablet; Drug: FM101 oral solution
- Phase 2a (Experimental)
  Interventions: Drug: Placebo; Drug: FM101 150 mg; Drug: FM101 300 mg

INTERVENTIONS:
Drug: FM101 tablet — Bio-equivalent test (tablet vs oral solution)
  Arms: Bioequivalent test of FM101 oral solution and FM101 tablet
Drug: FM101 oral solution — Bio-equivalent test (tablet vs oral solution)
  Arms: Bioequivalent test of FM101 oral solution and FM101 tablet
Drug: Placebo — Placebo BID for 28 days
  Arms: Phase 2a
Drug: FM101 150 mg — FM101 (150 mg) BID for 28 days
  Arms: Phase 2a
Drug: FM101 300 mg — FM101 (300 mg) BID for 28 days
  Arms: Phase 2a

SUMMARY:
A PHASE 1/2A, RANDOMIZED, DOUBLE-MASKED, PLACEBO-CONTROLLED, MULTI-CENTER STUDY ASSESSING THE SAFETY, TOLERABILITY, AND EFFICACY OF FM101 IN PATIENTS WITH OCULAR HYPERTENSION, AND TO ASSESS THE RELATIVE BIOAVAILABILITY OF THE FM101 ORAL TABLET FORMULATION IN HEALTHY PARTICIPANTS

ELIGIBILITY:
Inclusion Criteria:

* Sex : Male or female patients.
* Age : 18 to 75 years, inclusive, at screening.
* BMI : 18.0 to 32.0 kg/m2.
* Weight : ≥50 kg.
* Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or use highly effective contraceptive method (oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones, a vaginal ring or an intrauterine device [IUD]) from screening until study completion, including the follow-up period for at least 90 days after the last dose of study drug, or be post-menopausal for ≥12 months. Post-menopausal status will be confirmed through testing of FSH levels (≥30 IU/mL) at screening for amenorrheic female participants. Females who are abstinent from heterosexual intercourse will also be eligible.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at screening and admission and be willing to have additional pregnancy tests as required throughout the study.
* Males must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, the participant and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from screening until study completion, including the follow-up period, for at least 90 days after the last dose of study drug. Male participants whose female partner is post-menopausal, and participants who are abstinent from heterosexual intercourse will also be eligible. Male participants must agree to refrain from donating sperm from screening until study completion, including the follow-up period, for at least 90 days after the last dose of study drug.
* Willing and able to participate in the study, give written informed consent, and comply with the study procedures.
* Diagnosis of OHT in at least 1 eye, not currently receiving medication for raised IOP or able to stop such medication for a washout period and the duration of the study.
* Elevated IOP (≥24 and ≤32 mmHg at 08:00 hours, and ≥21 and ≤32 mmHg at 12:00 hours) on baseline visit in at least one eye off treatment.
* Anterior chamber is open and non-occludable (both eyes) as confirmed by Investigator by gonioscopy examination at screening.

Exclusion Criteria:

* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at screening that the Investigator judges as likely to interfere with the objectives of the trial or the safety of the patient.
* Female patients who are pregnant, nursing, or planning a pregnancy. The absence of pregnancy will be confirmed for all female patients by a serum pregnancy test conducted at screening, and a urine pregnancy test on Day -1 and at follow-up.
* Patients with known or suspected drug or alcohol abuse.
* Current enrollment or past participation within the last 30 days before the screening visit in any other clinical study involving an investigational study treatment or any type of medical research.
* Patients with a history of poor study drug compliance, protocol non-compliance, or prohibited medication intake.
* Patients with a history or presence of uncontrolled, chronic, generalized, systemic, or other disease that the Investigator feels might increase the risk to the safety of the patient or confound the results of the study.
* Surgery (e.g., stomach bypass) or medical condition that might significantly affect absorption of medicines (as judged by the Investigator).
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
* Patients requiring concomitant medication (either systemic or topical) known to affect IOP (e.g., beta-blockers, calcium channel blockers, ACE inhibitors, CAIs, or corticosteroids). However, systemic antihypertensive medications are allowed as long as the dose and regimen have been stable for at least 3 months prior to screening and are expected to remain stable throughout the study.
* Receiving more than one medication for IOP at time of screening.
* Patients who used inhibitors or inducers of cytochrome P450 3A4 in the last 30 days.
* Uncontrolled intraocular hypertension in any eye defined as >30 mmHg at either of the screening/baseline visits (after a washout phase in those patients who were currently receiving ocular hypotensive therapy).
* Central corneal thickness of less than 500 µm or greater than 620 µm.
* BCVA worse than 20/200 in either eye.
* Any corneal abnormality or other condition interfering or preventing reliable Goldmann applanation tonometry (e.g., Fuchs dystrophy or significant corneal surface abnormality).
* Advanced glaucoma (e.g., cup/disc ratio >0.80), evidence of significant visual field defect that would be at risk for progression during the wait/washout period, or progressive visual field loss within the last year.
* Any other forms of glaucoma (e.g angle closure glaucoma, normal tension glaucoma, congenital glaucoma, etc), other than OAG or OHT.
* Use of contact lenses within one week prior to Day 1 until end of treatment.
* Patients with history of severe ocular trauma in either eye.
* Previous complicated surgery or glaucoma surgery or laser treatment of any kind in either eye.
* Presence of any active severe external ocular disease, inflammation, or infection of the eye and/or eyelids.
* History of retinal detachment, proliferative diabetic retinopathy, or any retinal disease that may be progressive during the time course of the study.
* Presence of clinically significant macular edema.
* Any ocular disease or condition that in the opinion of the study Investigator may put the patient at significant risk, may confound study results, or may interfere significantly with the patient's participation in the study.
* Donation or loss of more than 450 mL blood during the 3 months before the start of screening.
* Known allergy, hypersensitivity, or contraindications to FM101.
* Positive screen for HBsAg, HCV antibodies, or anti-HIV 1 and 2 antibodies.
* Any other condition that would confound the study or endanger the safety of the patient as per the judgment of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of two dose levels of FM101 after repeated dosing in patients with OAG or OHT compared to that of placebo. | Day 1 through Day 37
  The number of TEAEs (frequency of occurrence, number of subjects experiencing the event)
To assess the effect of two dose levels of FM101 in oral tablet formulation on the change from baseline intraocular pressure (IOP) in the study eye at 08:00 hours, after 28 days of repeated dosing in patients with OHT compared to that of placebo. | Day 1 through Day 28
  IOP change in the study eye at 8:00 from Baseline to Day 28
To assess the effect of two dose levels of FM101 in oral tablet formulation on the change from baseline intraocular pressure (IOP) in the study eye at 12:00 hours, after 28 days of repeated dosing in patients with OHT compared to that of placebo. | Day 1 through Day 28
  IOP change in the study eye at 12:00 from Baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jung Chul Kwon, Study Chair — Futuremedicine Australia Pty Ltd
Locations (5):
- Australia (5):
  - Norwest Eye Medical Pty Ltd, Bella Vista, New South Wales
  - Adelaide Eye & Retina Centre, Adelaide
  - CMAX Clinical Research Pty Ltd, Adelaide
  - Eye Surgery Associates, East Melbourne
  - Lions Eye Institute, Nedlands